CLINICAL TRIAL: NCT03195894
Title: Clinical Study of TripleA Connected to Diagnosis, Care and Aftercare of Alcohol Addiction in Outpatient Care
Brief Title: Clinical Study of TripleA for Treatment of Alcohol Addiction in Outpatient Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kontigo Care AB (Industry)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: KC102-001/KC102-002
Record Dates: First submitted 2017-05-11; First posted 2017-06-22 (Actual); Results first posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Alcoholism
Keywords: Alcohol abuse, Alcoholometer, Medical Device, App
MeSH Terms: conditions — Alcoholism; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, open study to compare conventional treatment with and without addition of TripleA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment and TripleA (Experimental): Conventional treatment and TripleA medical device consisting of alcoholometer, a Bluetooth mobile app on cell phone and information stored on computer for caregiver
  Interventions: Device: TripleA
- Conventional treatment (No Intervention): Conventional treatment

INTERVENTIONS:
Device: TripleA
  Arms: Conventional treatment and TripleA

SUMMARY:
The primary objective is to investigate differences in the alcohol consumption pattern between alcohol addicts receiving conventional treatment and those who receive a combination of conventional treatment and TripleA.

DETAILED DESCRIPTION:
The study is a 12-month open-label and randomised comparison between the control group receiving only conventional treatment and the intervention group receiving conventional treatment enhanced with TripleA.

The studies have been designed to reflect as far as possible the conventional care for alcohol dependence. The TripleA product is intended to strengthen the existing methods used during the assessment phase, treatment phase and aftercare of alcohol dependence.

ELIGIBILITY:
Inclusion Criteria:

* Patients in care at Addiction and Neuropsychiatry Uppsala University Hospital and at Nämndemansgården Uppsala
* 18 years or older
* Meets at least 2 of the criteria for addiction/substance syndrome according to Diagnostic and statistical manual of mental disorders-5 (DSM-5)
* Ability to understand and communicate in Swedish
* Ability to handle the technical equipment used in the study (alcoholometer and Smartphone)
* Access to a fixed place (living, place for sleeping, place where the phone can be charged

Exclusion Criteria:

* Schizophrenia
* Substance syndrome related to other substances than alcohol and nicotin
* Lowered lung function (not able to reach acceptable expiration volume for the alcoholometer function)
* The patient is taken care of within the frame for The Act on Care of Addicts
* Not suitable to participate according to the Investigator
* Has not consumed any alcohol during the 4 weeks defined as baseline timeline follow back
* Normalized Carbohydrate Deficient Transferrin (CDT) and Phosphatidyl-Ethanol (PEth)-values in blood samples at visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Eriksson, MD PhD, Principal Investigator — Uppsala University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamalainen MD, Zetterstrom A, Winkvist M, Soderquist M, Karlberg E, Ohagen P, Andersson K, Nyberg F. Real-time Monitoring using a breathalyzer-based eHealth system can identify lapse/relapse patterns in alcohol use disorder Patients. Alcohol Alcohol. 2018 Jul 1;53(4):368-375. doi: 10.1093/alcalc/agy011. PMID 29590325

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at two sites (Uppsala University Hospital and Nämndemansgården) beginning in October 2015 . Recruitment continued until January 2017 and the last follow-up visits were conducted in December 2017 (Uppsala University Hospital) and in January 2018 (Nämndemansgården), respectively.
Groups:
- Conventional Treatment: Conventional treatment may be medication or 12-step addiction treatment according to the Minnesota model.
Period: Overall Study
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Started | 59 | 56
Completed | 26 | 28
Not Completed | 33 | 28
Not completed — An example is "Started other treatment". | 4 | 5
Not completed — Withdrawal by Subject | 15 | 4
Not completed — Lost to Follow-up | 14 | 19

BASELINE CHARACTERISTICS:
Population: Patients (n=115) were recruited to clinical trials from a 12-step aftercare programme(12S-ABS) and from hospital care with abstinence (HC-ABS) or controlled drinking (HC-CDR) as goal. The subject population for study KC102-001 was formed by 71 subjects enrolled at Uppsala University Hospital. Study KC102-002 included 44 subjects registered at Nämndemansgårdens treatment home.
Groups:
- Conventional Treatment and TripleA: Conventional treatment and TripleA medical device consisting of alcoholometer, a Bluetooth mobile app on cell phone and information stored on computer for caregiver TripleA.
- Conventional Treatment: Conventional treatment which is medication or a 12-step addiction treatment according to the Minnesota model.
- Total: Total of all reporting groups
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment | Total
Number analyzed (Participants) | 59 | 56 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (8.16) | 53.8 (9.63) | 53.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 39
  Male | 37 | 39 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 59 | 56 | 115

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With no Heavy Drinking Days After 12 Months
Description: Difference between the treatment arms in percentage of patients with no heavy drinking days during the 4-weeks period before the 12 months follow-up visit .
Time Frame: Four weeks period before the 12 months visit
Population: Of the planned patient number (216 patients) only approximately 25% or less was analyzed due to poor recruitment rate and a high drop-out of patients during the study.
Measure: Count of Participants; unit: Participants
Groups:
- Conventional Treatment: Conventional treatment only.
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 26 | 28
Participants | 8 | 9

2. Secondary Outcome: Percentage of Sober Patients During the Period Before the 6 Months Visit
Description: Difference in percentage of sober patients (zero drinks during one month reporting period) during the four weeks period before the 6 months visit.
Time Frame: The four weeks-period before the 6 months visit
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 38 | 37
Participants | 24 | 21

3. Secondary Outcome: Percentage of Sober Patients Before the 12 Months Visit
Description: Percentage of sober patients (zero drinks during one month reporting period) during the four weeks period before the 12 months visit.
Time Frame: The four weeks-period before the 12 months visit
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 26 | 28
Participants | 15 | 14

4. Secondary Outcome: Change in Total Amount of Consumed Alcohol From the Baseline Visit to the 6 Months Visit
Description: Number of drinks during the 4 weeks period before the baseline visit minus number of drinks during the 4 weeks period before the 6 months visit. A positive difference means a reduction in drinking. A negative difference means increased drinking.
Time Frame: The four weeks-period before the baseline visit and before the 6 months visit
Measure: Mean (Standard Deviation); unit: Number of drinks
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 38 | 37
Number of drinks | 183.7 (147.27) | 180.62 (187.91)

5. Secondary Outcome: Change in Total Amount of Consumed Alcohol From the Baseline Visit to the12 Months Visit
Description: Number of drinks during the 4 weeks period before the baseline visit minus number of drinks during the 4 weeks period before the 12 months visit. A positive difference means a reduction in drinking. A negative difference means increased drinking.
Time Frame: The four weeks-period before the baseline visit and before the 12 months visit
Measure: Mean (Standard Deviation); unit: Number of drinks
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 26 | 28
Number of drinks | 195.02 (170.29) | 150.93 (164.09)

6. Secondary Outcome: Change in Heavy Alcohol Drinking Days From the Baseline Visit to the 6 Months Visit
Description: Number of heavy drinking days during the 4 weeks period before the baseline visit minus number of heavy drinking days during the 4 weeks period before the 6 months visit. A positive difference means a reduction in drinking. A negative difference means increased drinking.
Time Frame: The four weeks-period before the baseline visit and before the 6 months visit
Measure: Mean (Standard Deviation); unit: Number of heavy drinking days
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 38 | 37
Number of heavy drinking days | 15.21 (10.79) | 14.41 (10.02)

7. Secondary Outcome: Change in Heavy Alcohol Drinking Days From the Baseline Visit to the 12 Months Visit
Description: Number of heavy drinking days during the 4 weeks period before the baseline visit minus number of heavy drinking days during the 4 weeks period before the 12 months visit. A positive difference means a reduction in drinking. A negative difference means increased drinking.
Time Frame: The four weeks-period before the baseline visit and before the 12 months visit
Measure: Mean (Standard Deviation); unit: Number of heavy drinking days
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 26 | 28
Number of heavy drinking days | 14.65 (10.61) | 13.54 (10.23)

8. Secondary Outcome: Change in Number of Sober Days Before the Baseline Visit Compared to the 6 Months Visit
Description: Number of sober days during the 4 weeks period before the baseline visit minus number of sober days during the 4 weeks period before the 6 months visit. A negative difference means a reduction in drinking. A positive difference means increased drinking.
Time Frame: The four weeks-period before the baseline visit and before the 6 months visit
Measure: Mean (Standard Deviation); unit: Difference in number of sober days
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 38 | 37
Difference in number of sober days | -15.87 (10.11) | -15.35 (10.58)

9. Secondary Outcome: Change in Number of Sober Days Before the Baseline Visit Compared to Before the 12 Months Visit
Description: Number of sober days during the 4 weeks period before the baseline visit minus number of sober days during the 4 weeks period before the 12 months visit. A negative difference means a reduction in drinking. A positive difference means increased drinking.
Time Frame: The four weeks-period before the baseline visit and before the 12 months visit
Measure: Mean (Standard Deviation); unit: Difference in number of sober days
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 26 | 28
Difference in number of sober days | -14.38 (9.80) | -13.04 (11.97)

10. Secondary Outcome: Change in Number of Standard Glasses Per Drinking Day Before the Baseline Visit Compared to Before the 6 Months Visit
Description: Number of standard glasses/drinks per drinking day during the 4 weeks period before the baseline visit minus number of standard glasses/drinks per drinking day during the 4 weeks period before the 6 months visit. A positive difference means a reduction in drinking. A negative difference means increased drinking.
Time Frame: The four weeks-period before the baseline visit and before the 6 months visit
Measure: Mean (Standard Deviation); unit: Average no of glasses per drinking day
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 38 | 37
Average no of glasses per drinking day | 7.70 (5.73) | 7.36 (7.62)

11. Secondary Outcome: Change in Number of Standard Glasses Before the Baseline Visit Comapred to Before the 12 Months Visit
Description: Number of standard glasses/drinks per drinking day during the 4 weeks period before the baseline visit minus number of standard glasses/drinks per drinking day during the 4 weeks period before the 12 months visit. A positive difference means a reduction in drinking. A negative difference means increased drinking.
Time Frame: The four weeks-period before the baseline visit and before the 12 months visit
Measure: Mean (Standard Deviation); unit: Average no of glasses per drinking day
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 26 | 28
Average no of glasses per drinking day | 8.52 (6.61) | 7.03 (6.37)

12. Secondary Outcome: Time to Heavy Drinking
Description: Time period in days from randomization to first heavy drinking day. Longer time means a better result.
Time Frame: From date of randomization until the date of first heavy drinking day, assessed up to 12 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 59 | 56
Days | 187.3 (139.3) | 141.2 (134.6)

13. Secondary Outcome: Change in Health Outcome, Measured With the Visual Analog Scale (EQ VAS) in EQ-5D at the Baseline Visit Compared to the 6 Months Visit
Description: Change in health outcome, measured with the visual analog scale (EQ VAS) in EQ-5D after 6 months compared to baseline. The EQ-5D is a standardized instrument for measuring and describing health outcomes. VAS score is 0-100 where 0 is the worst possible health and 100 is the best possible health. A positive difference indicates improvement.
Time Frame: Baseline, After 6 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 37 | 37
Score on a scale | 9.84 (21.52) | 6.27 (22.28)

14. Secondary Outcome: Change in Health Outcome, Measured With the Visual Analog Scale (EQ VAS) in EQ-5D From the Baseline Visit Compared to the 12 Months Visit
Description: Change in health outcome, measured with the visual analog scale (EQ VAS) in EQ-5D after12 months compared to baseline. The EQ-5D is a standardized instrument for measuring and describing health outcomes. VAS score is 0-100 where 0 is the worst possible health and 100 is the best possible health. A positive number indicates improvement.
Time Frame: Baseline, After 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 26 | 28
score on a scale | 6.23 (22.07) | 8.18 (20.43)

15. Secondary Outcome: Change in Health Outcome Measured With the Questionnaire in EQ5D After 6 Months Compared to Baseline
Description: Change in health outcome, measured with the questionnaire in EQ-5D after 6 months compared to baseline. The questionnaire EQ-5D in EQ-5D consists of 5 questions giving score 5 - 15. A higher positive number indicates improvement.
Time Frame: Baseline, After 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 38 | 37
score on a scale | 0.16 (1.41) | 0.08 (1.12)

16. Secondary Outcome: Change in Health Outcome, Measured With the Questionnaire in EQ-5D After 12 Months Compared to Baseline
Description: Change in health outcome, measured with the questionnaire in EQ-5D after 12 months minus baseline. The questionnaire EQ-5D in EQ-5D consists of 5 questions giving score 5 - 15. A higher positive number indicates improvement.
Time Frame: Baseline, After 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 26 | 28
score on a scale | -0.04 (1.37) | 0.32 (0.98)

17. Secondary Outcome: Percentage of Patients Who Have Reduced Their AUDIT Score After 12 Months
Description: Percentage of patients who have reduced their AUDIT score (Alcohol Use Disorders Identification Test, score 0-40) after 12 months. Higher proportion is better.
Time Frame: After 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 25 | 28
Participants | 24 | 24

18. Secondary Outcome: Percentage of Patients With Lowered AUDIT Score With at Least One Zone After 12 Months
Description: Percentage of patients who have reduced their Alcohol Use Disorders Identification Test (AUDIT) risk zones with at least one zone. Higher proportion is better.
Time Frame: After 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 25 | 28
Participants | 21 | 23

19. Secondary Outcome: Percentage of Patients Having a Risk Level <II (i.e. Less Than 6 AUDIT Points for Women, 8 AUDIT Points for Men) After 12 Months
Description: Percentage of patients having a risk level <II (i.e. less than Alcohol Use Disorders Identification Test (AUDIT) points, i.e. 6 points for women, 8 points for men) after 12 months. Higher proportion is better.
Time Frame: After 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 26 | 28
Participants | 13 | 9

20. Secondary Outcome: Change in Degree of Alcohol Dependence Measured as the Difference in SADD-points at Baseline Compared to 6 Months
Description: Change in degree of alcohol dependence measured as the difference in Short Alcohol Dependence Data (SADD)-points at baseline minus 6 months Scoring: The 15 items summed for a total score than can range from 0 to 45. Scale totals are interpreted as follows: 1-9 low dependence, 10-19 medium dependence, and 20 or greater high dependence. A large positive number indicates a better result.
Time Frame: Baseline, After 6 months
Measure: Mean (Standard Deviation); unit: Difference in SADD-points
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 38 | 37
Difference in SADD-points | 15.39 (9.53) | 11.76 (9.60)

21. Secondary Outcome: Change in Degree of Alcohol Dependence Measured as the Difference in SADD-points at Baseline Compared to 12 Months
Description: Change in degree of alcohol dependence measured as the difference in Short Alcohol Dependence Data (SADD)-points at baseline minus 12 months. Scoring: The 15 items summed for a total score than can range from 0 to 45. Scale totals are interpreted as follows: 1-9 low dependence, 10-19 medium dependence, and 20 or greater high dependence. A large positive number indicates a better result.
Time Frame: Baseline, After 12 months
Measure: Mean (Standard Deviation); unit: Difference in SADD-points
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 26 | 27
Difference in SADD-points | 17.00 (10.56) | 11.19 (9.17)

22. Secondary Outcome: Compliance With Agreed Treatment
Description: Percentage of subjects staying in the study to the 12 months visit.
Time Frame: Baseline, After 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 59 | 56
Participants | 26 | 28

23. Secondary Outcome: Change in Concentration of the Alcohol Metabolite PEth at Baseline Compared to 6 Months Visit
Description: Change in concentration of the alcohol metabolite PEth at baseline minus 6 months. A larger positive change of PEth concentration is a better outcome.
Time Frame: Baseline, After 6 months
Measure: Mean (Standard Deviation); unit: umol/L
Groups:
- Conventional Treatment: Conventional treatment consisting of medication treatment or the Minnesota model of addiction treatment
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 18 | 29
umol/L | 0.20 (0.61) | 0.33 (0.85)

24. Secondary Outcome: Change in Concentration of the Alcohol Metabolite PEth at Baseline Compared to 12 Months
Description: Change in concentration of the alcohol metabolite PEth at baseline minus 12 months. A larger positive change of PEth concentration is a better outcome.
Time Frame: Baseline, After 12 months
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 12 | 25
umol/L | 0.53 (0.86) | 0.18 (0.37)

25. Secondary Outcome: Change in Concentration of the Alcohol Metabolite CDT in the Blood at Baseline Compared to 6 Months
Description: CDT (Carbohydrate Deficient Transferrin) concentration is given in % of total transferrin in serum, i e. CDT(%). The change is calculated as baseline CDT (%) minus CDT(%) at 6 months. A large positive difference indicates decreased drinking.
Time Frame: Baseline, After 6 months
Measure: Mean (Standard Deviation); unit: percentage CDT of total transferrin
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 12 | 19
percentage CDT of total transferrin | 0.11 (0.55) | 0.42 (0.94)

26. Secondary Outcome: Change in Concentration of the Alcohol Metabolite CDT in the Blood at Baseline Compared to 12 Months
Description: CDT (Carbohydrate Deficient Transferrin) concentration is given in % of total transferrin in serum, i e. CDT(%). The change is calculated as baseline CDT (%) minus CDT(%) at 12 months. A large positive difference indicates decreased drinking.
Time Frame: Baseline, After 12 months
Measure: Mean (Standard Deviation); unit: percentage CDT of total transferrin
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
Number analyzed (Participants) | 8 | 16
percentage CDT of total transferrin | 0.18 (0.70) | 0.25 (0.74)

ADVERSE EVENTS:
Time Frame: Safety with collection of adverse events was followed for each patient from Baseline (start of study) until the 12-month visit (end of study).
Arm/Group | Conventional Treatment and TripleA | Conventional Treatment
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/56
Serious Adverse Events (participants affected / at risk) | 12/59 | 6/56
Other Adverse Events (participants affected / at risk) | 5/59 | 4/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Treatment and TripleA (N=59) | Conventional Treatment (N=56)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) — Ascites due to liver cirrhosis. Not related to device.
Bleeding (Gastrointestinal disorders) | 1 (2) | 0 (0) — Bleeding esophagusvarices and duodenal ulcus. Not related to device.
Sepsis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Staphylococcus aureus sepsis. Not related to device.
Abstinence (Psychiatric disorders) | 6 (9) | 2 (2) — Hospitalization due to alcohol abstinence. Not related to device.
Fainting, dizziness and nausea (General disorders) | 1 (1) | 1 (1) — Not related to device.
Suspected transient ischemic attack (TIA) (Vascular disorders) | 0 (0) | 1 (1) — Not related to device.
Infection in foot (Infections and infestations) | 0 (0) | 1 (1) — Infection in foot after surgery. Not related to device.
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Not related to device.
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) — Not related to device.
Alcohol intoxication (General disorders) | 2 (2) | 0 (0) — Intoxication, lowered consciousness and delirium. Not related to device.
Suicide attempts (Psychiatric disorders) | 1 (1) | 0 (0) — Not related to device.
Recurrent ischemic pain (Vascular disorders) | 1 (1) | 0 (0) — Not related to device
Myocardial Infarction (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Treatment and TripleA (N=59) | Conventional Treatment (N=56)
Cold, fever, flu (Infections and infestations) | 2 (3) | 3 (3) — Five patients reported cold, or flu-like symptoms and fever.
Pain (General disorders) | 3 (3) | 1 (1) — Four patients reported pain in foot, hand, or thumb.

LIMITATIONS AND CAVEATS:
Due to unrealistic assumptions in the sample size calculations, difficulties in recruiting subjects and high dropout rate, the study was inconclusive.

The poor recruitment rate and poor retention of patients in the study was a challenge (in addition with the quality of self-reported outcomes). The drop-out rate, especially between month 6-12, was a problem both in treatment and control groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT03195894/Prot_SAP_000.pdf